CLINICAL TRIAL: NCT05828212
Title: A Study on the Safety and Efficacy of Chimeric Antigen Receptor T Cells in the Treatment of Recurrent/Refractory Neuromyelitis Optica
Brief Title: Evaluate the Safety and Efficacy of CAR-T Cells in the Treatment of R/R Neuromyelitis Optica
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2023005
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Recurrent/Refractory Neuromyelitis Optica
  Interventions: Drug: CAR-T cells injection

INTERVENTIONS:
Drug: CAR-T cells injection — CAR-T cells in the treatment of R/R neuromyelitis optica

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD19 CAR-T therapy for patients with relapsed or refractory Neuromyelitis Optica, and to evaluate the pharmacokinetics of CD19 CAR-T in patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-60 and gender unlimited;
* 2. NMOSD diagnosed based on the 2015 NMOSD International Consensus Diagnostic Criteria;
* 3. Diagnostic criteria for AQP4-IgG positive NMOSD Diagnostic criteria for AQP4-IgG positive NMOSD

  1. At least 1 core clinical feature
  2. Using reliable methods to detect positive AQP4-IgG (CBA method)
  3. Exclude other diagnoses. Core clinical features

  <!-- -->

  1. ＯＮ
  2. Acute myelitis
  3. Posterior region syndrome, unexplained paroxysmal hiccup, nausea, and vomiting
  4. Other brainstem syndromes
  5. Symptomatic episodic sleeping sickness, diencephalic syndrome, brain MRI with NMOSD characteristic diencephalic lesions
  6. Cerebral syndrome with NMOSD characteristic brain lesions
* 4. Corticosteroids combined with immunosuppressants (azathioprine or mycophenolate mofetil or rituximab) still relapse after treatment；
* 5. At least 2 relapses within the past 12 months or at least 3 relapses within the past 24 months, and at least 1 recurrence within the 12 months prior to screening；
* 6. The estimated survival time is more than 12 weeks;
* 7. Women of childbearing age who have negative urine pregnancy test before medication administration and agree to take effective contraceptive measures during the trial period until the last follow-up

Exclusion Criteria:

* 1. Epilepsy history or other central nervous system disease;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythm ia in the past;
* 3. Pregnant (or lactating) women;
* 4. Patients with severe active infections;
* 5. Active infection of hepatitis B virus or hepatitis C virus;
* 6. Systemic steroids have used in the 4 weeks before participating in the treatment (except recently or currently using inhaled steroids);
* 7. Those who have used any gene therapy products before;
* 8. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 9. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
* 10. Those who suffer from other uncontrolled diseases are not suitable to join the study;
* 11. HIV infection;
* 12. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | From date of initial treatment to Day 28 post CAR-T infusion.
  Dose limited toxicity
AE and SAE | From admission to the end of the follow-up, up to 2 years
  Adverse event and serious adverse event
Maximum tolerable dose | From date of initial treatment to Day 28 post CAR-T infusion.
  Maximum tolerable dose

SECONDARY OUTCOMES:
Changes in serum AQP4-IgG titer after infusion | days 7, 14, 21, 28 and 90
  Changes in serum AQP4-IgG titer after infusion
Annual recurrence rate (ARR) of NMOSD | From admission to the end of the follow-up, up to 2 years
  Annual recurrence rate (ARR) of NMOSD
Changes in the expanded disability status scale (EDSS) score from baseline | days 7, 14, 21, 28 ,56 and 90
  EDSS:0 (normal neurological exam) to 10 (death due to MS),Higher scores indicate greater disability (worse outcome)，Score reduction suggests functional improvement
MRI active lesions | days 90
  Proportion of subjects with ≥1 active lesions at Day 90
Changes in optimal corrected vision | days 28 and 90
  Changes in optimal corrected vision (Log MAR)
Changes of nerve fiber layer around the retinal papilla(pRNFL) | 2 years
  Change in RNFL by optical coherence tomography over trial
Changes in the plexiform layer of macular ganglion cells (mGCIPL) | 2 years
  Proportion of subjects with significant mGCIPL thickness changes

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China